CLINICAL TRIAL: NCT01429324
Title: Validation of Near Infrared Spectroscopy (NIRS) Neuro-monitoring During Deep Hypothermic Circulatory Arrest for Aortic Arch Surgery
Brief Title: Near Infrared Spectroscopy (NIRS)
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: Mod11-000295-03
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Aortic Arch Surgery
Keywords: Near infrared spectroscopy; neuromonitoring; aortic arch surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac disease: Aortic arch surgery

SUMMARY:
This study is designed to assess the feasibility of evaluating cerebral saturation during critical periods of deep hypothermia circulatory arrest and Selective Antegrade Cerebral Perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female
* Is of any race or ethnicity
* Is greater than or equal to eighteen (18) years of age
* Weighs greater than or equal to 40 kilogram
* Is not known to be pregnant
* Understands English
* Is undergoing aortic arch surgery with planned deep hypothermia circulatory arrest, either with or without select antegrade cerebral perfusion
* Is able and willing to provide informed consent

Exclusion Criteria:

* Is less than eighteen (18) years of age
* Weighs less than 40 kilogram
* Is known to be pregnant
* Does not understand English
* Has known sensitivity to adhesives
* Is unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic and affiliated hospitals
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evaluate brain tissue oxygenation assessing the number and percentage of subjects from whom regional data could be collected during 90% of the aortic arch surgery, and the registration rate during deep hypothermic circulatory arrest. | At the end of the surgical case approximately 6 to 8 hours

SECONDARY OUTCOMES:
Determine whether there are unilateral or global differences in cerebral tissue oxygenation detected during selective antegrade cerebral perfusion | At the end of the surgical case approximately 6 to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: James J Lynch, MD, Principal Investigator — Mayo Clinic and affiliated hospitals
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States